CLINICAL TRIAL: NCT02346162
Title: PREPARE: A Randomized Trial of a Pre-pregnancy Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DK099882 (NIH); R01DK099882 (NIH)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Overweight; Obese
Keywords: Pre-pregnancy; Weight management
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Weight management intervention
  Interventions: Behavioral: Weight management
- Usual Care Control (Other): Usual Care for planning healthy pregnancy
  Interventions: Other: Usual Care Control

INTERVENTIONS:
Behavioral: Weight management — Phone counseling for pre-pregnancy weight loss and weight maintenance when BMI </=25, and when pregnant, weight gain within IOM guidelines.
  Arms: Intervention
Other: Usual Care Control — Usual care control participants receive general dietary advice as it relates to planning for a healthy pregnancy (e.g. folate requirements, prenatal vitamins, smoking cessation, alcohol cessation, and prenatal food safety).
  Arms: Usual Care Control

SUMMARY:
The US obesity epidemic is being transmitted to the next generation. Growing evidence suggests that both a mothers' weight at pregnancy onset, and excessive weight gain during pregnancy, are associated with increased risk of pregnancy-related complications such as gestational diabetes and pre-eclampsia, and an increased risk that her child will become obese and face obesity-related health issues in later life.

Currently, over one-third of reproductive-aged women in the U.S. are obese [body mass index (BMI) ≥ 30]. Our research team has shown that we can improve birth weight outcomes in babies of obese women who start a weight-management intervention program at 14 to 15 weeks of their pregnancy (soon after their first prenatal visit). However, organogenesis and metabolic programming begin early in the first trimester, well before the first prenatal visit. Therefore, waiting to address mothers' weight, physical activity, and diet quality until the first prenatal visit is not optimal. Given the need to reach overweight and obese women prior to pregnancy, and the Institute of Medicine's (IOM's) recent recommendation, based on observational studies, that women should reach a healthy weight before conceiving, this randomized clinical trial will evaluate a comprehensive preconception weight loss program.

DETAILED DESCRIPTION:
The goals are to help overweight and obese women (BMI ≥ 27) who are considering pregnancy to adopt improved dietary and physical activity habits and lose weight prior to becoming pregnant, and then help them maintain those habits and prevent excessive weight gain during their pregnancy. We model this intervention after successful, frequent-contact interventions designed by ourselves and other investigators. We start with face-to-face counseling followed by frequent telephone counseling contacts. The expected outcomes for mothers include reduced pregnancy-related weight gain (primary) and lower weight at the start of pregnancy (secondary) and for babies, decreased risk of exceeding national norms for weight at birth (secondary).

ELIGIBILITY:
Inclusion Criteria:

* Current Kaiser Permanente Northwest (KPNW) member
* Expects to be KPNW member for at least 2 more years
* Body Mass Index (BMI) ≥ 27
* Not currently pregnant
* Access to computer with Internet
* Completion of screening diet assessment
* English speaking

Exclusion Criteria:

* Taking medication (insulin or pills) for treatment of diabetes
* Gastrointestinal disease requiring special diet or medications (for example, ulcerative colitis, celiac sprue, phenylketonuria)
* Currently receiving treatment for cancer
* Renal disease (kidney disease requiring special diet or medication)
* History of bariatric surgery
* Use of prescription weight loss medications in the last three months
* Another household member already participating in the Prepare study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2015-06; Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Reduced pregnancy-related weight gain | 1 day at the end of pregnancy

SECONDARY OUTCOMES:
Lower weight at the start of pregnancy | Self-reported pre-pregnancy weight supplemented by weight at first prenatal visit (1 day)
Decreased risk of exceeding national norms for weight at birth | birth

CONTACTS AND LOCATIONS:
Overall Officials: Erin S LeBlanc, MD, Principal Investigator — Center for Health Research, Kaiser Permanente Northwest; Victor J Stevens, PhD, Principal Investigator — Center for Health Research, Kaiser Permanente Northwest
Locations (1):
- Anna Edelmann, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Any information from this study we present in reports or publications will not identify any individual.

REFERENCES:
- [Result] LeBlanc ES, Smith NX, Vesco KK, Paul IM, Stevens VJ. Weight loss prior to pregnancy and subsequent gestational weight gain: Prepare, a randomized clinical trial. Am J Obstet Gynecol. 2021 Jan;224(1):99.e1-99.e14. doi: 10.1016/j.ajog.2020.07.027. Epub 2020 Jul 18. PMID 32687819
- [Derived] LeBlanc ES, Boisvert C, Catlin C, Lee MH, Smith N, Vesco KK, Savage J, Mitchell DC, Gruss I, Stevens VJ. Prepare randomized clinical trial: Acceptability, engagement, and lifestyle effects of a weight loss intervention beginning in pre-pregnancy. Obes Sci Pract. 2022 Feb 24;8(5):603-616. doi: 10.1002/osp4.596. eCollection 2022 Oct. PMID 36238226
- [Derived] LeBlanc ES, Smith NX, Vesco KK, Hillier TA, Stevens VJ. Weight Loss Prior to Pregnancy and Early Gestational Glycemia: Prepare, a Randomized Clinical Trial. J Clin Endocrinol Metab. 2021 Nov 19;106(12):e5001-e5010. doi: 10.1210/clinem/dgab547. PMID 34313765